CLINICAL TRIAL: NCT02355834
Title: Improving Continence in People With Inflammatory Bowel Disease: Active Case Finding and a Randomised Controlled Trial
Brief Title: Faecal Incontinence iNtervention Study
Acronym: FINS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Collaborators: Queen Mary University of London (Other); King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RD14/042
Record Dates: First submitted 2014-12-12; First posted 2015-02-04 (Estimated); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Fecal Incontinence; Inflammatory Bowel Disease (IBD)
Keywords: Fecal Incontinence (FI); Inflammatory bowel disease (IBD); bowel control; Chronic diarrhoea; rectal inflammation
MeSH Terms: conditions — Fecal Incontinence; Inflammatory Bowel Diseases; Proctitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (IBD Nurse CONSULT + BOOKLET) (Experimental): IBD nurse intervention-Will have 3-4 x 30 minute face-to-face sessions over 3 months with an IBD specialist nurse specifically focusing on bowel control. Participants completing at least 3 sessions will be considered to have completed the intervention. They will also be given a booklet and access to all usual care, including nurse-led IBD helpline
  Interventions: Other: IBD nurse intervention
- Group 2 (BOOKLET alone) (No Intervention): Will receive the same booklet and access to usual care as Group 1.

INTERVENTIONS:
Other: IBD nurse intervention — Two IBD nurse specialists at each centre (8 in total) will deliver the IBD nurse intervention
  Arms: Group 1 (IBD Nurse CONSULT + BOOKLET)

SUMMARY:
Inflammatory Bowel Disease (IBD) affects 250,000 adults in the United Kingdom (UK) and causes bouts of diarrhoea which are hard to control. Over a quarter of patients experience extremely distressing faecal incontinence (FI). Even when the disease is in remission, the majority of patients live in fear of not finding a toilet in time. This curtails their activities and quality of life. The National Institute for Clinical Excellence (NICE 2007) has issued national guidance on actively asking patients about FI and a step-wise care plan for managing FI. However, this has not been evaluated in people with IBD, the vast majority of whom do not ask for help, even when they have frequent FI.

Across six expert centres in the UK, the investigators will perform 3 linked studies: [1] The investigators will screen people with IBD, offering the opportunity to obtain help with bowel control. The investigators will compare uptake of a postal approach versus response to a proactive face-to-face asking approach at a physical or telephone clinical appointment. [2] The investigators will conduct a randomised controlled trial (RCT) comparing two different approaches (IBD nurse specialist plus self-help booklet versus self-help booklet alone) to see which one produces the best results in terms of reductions in FI, other symptoms, costs and quality of life at 6 months after intervention. Booklet group participants may access the nurse intervention at 6 months if they wish, when the RCT is finished. [3] Interviews will be performed at the end of the intervention, gathering patient views and preferences and staff perspectives via Qualitative interviews and free text questionnaire comments, to enable a rich understanding and interpretation of our results.

The investigators will disseminate the results widely to people with IBD and health professionals and take active steps to embed successful interventions in NHS services, having gained sound evidence on how many people want help, whether intervention is effective in improving FI, and patient and staff views on interventions.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) affects approximately 250,000 UK adults. It causes symptoms including diarrhoea and extreme faecal urgency and has an unpredictable relapsing-remitting course. A quarter of people with IBD report faecal incontinence (FI) and two-thirds have urgency, even when IBD is in remission. Although this limits peoples' lives, most do not seek professional help. No study has determined whether nationally recommended approaches to FI would help people with IBD.

Research question Does implementation of the nationally (NICE)-recommended approach to active case-finding and step-wise management of FI improve bowel control and quality of life in people with IBD.

The investigators will address 3 objectives:

1. To implement 'active case finding' for FI and life-restricting faecal urgency in people with IBD, monitoring uptake of the offer of help and investigating barriers to accessing care.
2. To determine the effectiveness of implementing the algorithm of care proposed by NICE for people with FI in a randomised controlled trial compared to provision of the same information in a self-management booklet. The trial will measure the effects of each intervention at 6 months after completion of the intervention.
3. To obtain detailed qualitative feedback from patients and staff on the best way of enabling health-seeking, the experience of the intervention and suggestions for future service developments.

Plan of investigation We will conduct research in 6 UK specialist IBD services, in two phases with an integral qualitative element.

Phase 1: active case finding: will (a) Compare active case finding rates of disclosure for FI as recommended by NICE by using a postal, telephone or face to face approach; and (b) Determine currently unmet need for intervention for FI. All hospitals will conduct postal case-finding (1000 people) and all will conduct face to face or telephone questioning (1000 people) to compare numbers reporting FI and uptake of offer of intervention.

Phase 2: randomised controlled trial 186 patients with IBD and FI will be recruited (from people wanting help in Phase 1) to a parallel multicentre RCT comparing 2 interventions: (a) CONSULT + BOOKLET: 3-4 face to face or telephone consultations with an IBD specialist nurse who has received extra training on FI plus provision of a booklet developed with IBD patients on self-help for FI; (b) BOOKLET: intervention is booklet alone.

ELIGIBILITY:
For active case-finding: diagnosis of IBD,between 18 and 80 years of age; diagnosis of IBD confirmed with endoscopy / colonoscopy; no stoma.

For RCT and patient interviews: Patients with IBD who experience FI, are interested in interventions, and meet the following:

Inclusion criteria:

* Endoscopically confirmed IBD diagnosis
* Between 18 and 80 years of age
* No current flare-up of disease (self-report of usual symptoms when not in active flare)
* Reporting FI at least once in the past year
* With or without ileo-anal pouch plus:

Exclusion criteria:

* Under 18 or over 80
* Current disease flare-up (self-report of usual symptoms indicative of active flare)
* Course of specialist FI treatment in past year
* Previous major anal fistula surgery (surgical lay-open) or current perianal fistula
* Current stoma
* Current participation in another trial
* Inability to give informed consent (for example, due to reduced mental capacity)
* Inability to read or speak sufficient English to understand study documents, procedures and requirements

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2015-05; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
The St Mark's faecal incontinence score (0-24 scale) | At 6 months from recruitment
  Self-reported incontinence and protection (medications, use of incontinence pads) score. Four items are scored 0 - 4 (0 = never, 4 = daily) and three items are scored as 0 (No), or 2 or 4 (Yes). This yields an overall score of 0 - 24, a higher score indicating greater incontinence problems

SECONDARY OUTCOMES:
International Consultation on Incontinence - Inflammatory Bowel Disease (ICIQ-IBD) | At 6 months from recruitment
  Self-reported questionnaire. Participants provide an 'in remission' and / or an 'in relapse' score of 0 - 4 across 35 items in 3 domains: Domain A (IBD-FI symptoms) - 11 questions yield an overall score of 0 - 46; Domain B (IBD-FI Quality of Life) - the 14 questions yield an overall score of 0 - 56; Domain C (Other concerns) - the 10 questions yield an overall score of 0 - 42. In all domains, a higher score indicates worse symptoms, quality of life (QoL), or concerns. In each domain, subtracting the remission score from the relapse score reveals variation in symptoms, QoL and concerns between these two disease states. A higher variation score indicates greater fluctuation of these issues for the patient. This outcome measure has been developed by two of the study team and is being further tested / validated here.
Inflammatory Bowel Disease - Quality of Life (IBD-Q) | At 6 months from recruitment
  Self-reported IBD quality of life questionnaire. Respondents select one option from seven available, scored from 1 to 7 across 32 questions. This yields an overall score of 32 (high impact on quality of life) to 224 (low impact on quality of life. A higher overall score equals better quality of life. Responses can also be calculated across four different domains of: Bowel systems, emotional health, systemic systems, and social function, following instructions provided by the copyright holder.
Harvey Bradshaw Index (HBI) | At 6 months from recruitment
  Modified screening questionnaire to enable patient self-completion. Collects information about classic disease symptoms of Crohn's disease and extra-intestinal features. Scores of up to 4 indicate clinical remission, scores of 5 and over indicate relapse.
Simple Clinical Colitis Activity Index (SCCAI) | At 6 months from recruitment
  Modified screening questionnaire to enable patient self-completion. Collects information about classic disease symptoms of Ulcerative colitis and extra-intestinal features. Scores of up to 4 indicate clinical remission, scores of 5 and over indicate relapse.
Measure Yourself Medical Outcome Profile (MYMOP 2) | At 6 months from recruitment
  Participants set 2 goals for intervention, grading goals at baseline and then re-scoring after intervention, giving an individualised profile of the most bothersome symptom
European Quality of Life - 5 Dimensions (EQ-5D) | At 6 months from recruitment
  Self-reported quality of life [QoL] scale; participants indicate their current capabilities by selecting one of five options, across 5 domains: Mobility, Self-care, usual activities, pain or discomfort, and anxiety or depression. Option 1 is scored as '1' , option 5 is scored as '5'. This yields a total score of 5 - 25, a higher score indicating greater health problems. Respondents also indicate, on a 0-100 scale, how good or bad their health is on the day of completion. '0' = the worst health imaginable, whilst 100 = the best health imaginable.
The Brief Illness Perception Questionnaire (BIPQ) | At 6 months from recruitment
  The participant responds to eight questions about their condition, and the impact this has on them. Questions 1,2,5, 6 & 8 are scored 0 (no impact / effect) to 10 (Great impact / effect), yielding a total score of 0 - 50, a higher score indicates greater impact. Questions 3, 4 & 7 are scored 0 (no control, help from treatment or understanding) to 10 (great amount of control, help from treatment, and understanding) yielding a total score of 0 - 30, a lower score indicates worse control, help from treatment, and understanding. Finally, the participant identifies three factors which they believe to have contributed towards their health problem.
Study specific tool: Health economics | At 6 months from recruitment
  The participant reports interactions with health care professionals and investigative procedures (in addition to any required for the study), hospital visits / stays; any equipment, medication, travel or work-absence costs endured during the study period
Study-specific tool: Global perception of change | At 6 months from recruitment
  Participants report whether they feel their incontinence has got worse, stayed the same or improved. The also indicate which of the interventions offered to them via the study's self-management booklet were taken up, and how easy or difficult these were to comply with, or use. There is also an opportunity to provide free text responses about their experience of the intervention. Response options are not scored, and there is no overall score for this tool. It is used to assess the impact, usefulness and acceptability of the offered interventions, in order to inform future service delivery.
Medical record of escalation of treatment | Up to 6 months from recruitment
  Records changes (increases) in medical or surgical treatment during the course of the intervention as this may confound outcomes for the participant, or lead to withdrawal from the study.

CONTACTS AND LOCATIONS:
Overall Officials: Christine Norton, PhD, Principal Investigator — King's College London
Locations (6):
- United Kingdom (6):
  - St. Marks Hospital (London North West Healthcare NHS Trust), Harrow, London
  - Queen Elizabeth II Hospital, Kings Lynn, Norfolk
  - Bart's Health NHS Trust, London
  - Royal Free Hospital, London
  - Guy's & St Thomas' NHS Foundation Trust, London
  - John Radcliffe Hospital (Oxford University Hospitals NHS Trust), Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Norton C, Dibley LB, Hart A, Duncan J, Emmanuel A, Knowles CH, Stevens N, Terry H, Verjee A, Kerry S, Hounsome N. Faecal incontinence intervention study (FINS): self-management booklet information with or without nurse support to improve continence in people with inflammatory bowel disease: study protocol for a randomized controlled trial. Trials. 2015 Oct 6;16:444. doi: 10.1186/s13063-015-0962-0. PMID 26445224